CLINICAL TRIAL: NCT01380509
Title: To Compare the Relative Bioavailability of 375 mg Metronidazole Capsules (Kali) With That of Flagyl 375 mg Capsules( G.D. Searle, Inc) Under Fasting Conditions
Brief Title: Bioavailability Study of Metronidazole Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MTL-P2-155
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: To Determine the Bioequivalence Study Under Fasting
Keywords: Bioequivalence, single-dose, fasting
MeSH Terms: conditions — Fasting | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received kali product under fasting conditions
  Interventions: Drug: Metronidazole
- B (Active Comparator): Subjects received Searle product under fasting conditions
  Interventions: Drug: Flagyl

INTERVENTIONS:
Drug: Metronidazole — Capsules, single-dose, fasting
  Other Names: Flagyl Capsules
  Arms: A
Drug: Flagyl — Capsules, single-dose, fasting
  Other Names: Metronidazole Capsules
  Arms: B

SUMMARY:
The purpose of this study is to compare the single-dose Bioavailability of Kali and G.D. Searle, Inc.

DETAILED DESCRIPTION:
To compare the relative Bioavailability of Metronidazole 375 mg Capsules with that of Flagyl 375 mg Capsules in healthy, adult subjects under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all the following criteria may be included in the study
* Availability of subjects for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject.
* Males or females aged from 18 to 50 years with a body weight index (BMI) within 19-30; demographic data (sex, age, ethnic group, body weight, height and smoking habits) will be recorded and reported in the final report.
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance and must be recorded as such in the CRF (laboratory tests are presented in section 7.1.3)
* Healthy according to the laboratory results and physical examination
* Subjects should be non-or ex-smokers

Exclusion Criteria:

* Significant history of hypersensitivity to metronidazole or any related products as well as sever hypersensitivity reactions (like angioedema) to any drugs.
* Presence or history of significant gastrointestinal, liver or kidney disease,or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
* Females who are pregnant, lactating or are likely to become pregnant during the study periods.
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the study.
* Positive pregnancy test before or during the study.
* Presence or history of significant thyroid dysfunction (hypo or hyperthyroidism).
* Presence or history of significant hypoadrenalism.
* Presence or history of significant blood disorders (thrombocytopenia, hemophilia, bleeding, etc.).
* Presence or history of significant neurological disorders.
* Maintenance therapy with any drug, or significant history of drug dependency, alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic), or serious psychological disease.
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.).
* Participation in another clinical trial in the previous 28 days before day 1 of this study.
* Donation of 500mL of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 5 days before day 1 of this study.
* Positive urine screening of drugs of abuse (drug names are presented in section 7.1.4.).
* Positive results to HIV, HBsAg or anti-HCV tests.
* History of fainting upon blood sampling.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-08; Primary Completion 2002-09 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence
  To conclude bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sicard, M.D, Principal Investigator — Algotithme Pharma Inc
Locations (1):
- Algorithme Pharma, Laval, Quebec, Canada